CLINICAL TRIAL: NCT02398812
Title: The Interprofessional Medication Assessment for Older Patients - a Multicenter Randomized Trial in Primary Care Setting
Brief Title: The Interprofessional Medication Assessment for Older Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: East Savo Hospital District (Other)
Collaborators: University of Eastern Finland (Other); Finnish Medicines Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILMA
Record Dates: First submitted 2015-03-13; First posted 2015-03-26 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Multimorbidity; Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active comparator (Active Comparator): In addition to usual care, participants allocated to intervention group will receive medication assessment and treatment plan based on it
  Interventions: Other: Medication assessment and treatment plan based on it
- Usual care (No Intervention): Usual care (reference group).

INTERVENTIONS:
Other: Medication assessment and treatment plan based on it — Intervention
  * Phase I: A medication assessment conducted by an interprofessional team including nurse, pharmacist and physician. The assessment is based on current medication list and basic information cathered by nurse.
  * Phase II: This phase is needed if the assessment cannot be conducted safely without physical examination conducted by physician. The comprehensive interprofessional assessment takes place after the clinical examination conducted by home care physician.
  Arms: Active comparator

SUMMARY:
The objective of this pragmatic multi-center randomized controlled trial is to test the effectiveness of interprofessional medication assessment in older patients needing home care due to their diseases or decreased functional capacity in primary care. The main hypothesis is that intervention has a positive impact on functional capacity and for rational and safe use of medicines.

DETAILED DESCRIPTION:
Aging increases the risk of adverse effects and interactions caused by medication. Medication reconciliation and medication review are well-known practices to optimize medicines use. Both interventions usually require a team-based approach to be effective. Medication reconciliation is the process of obtaining and documenting a complete and accurate list of current patient medications and comparing this list with medication orders at each point of care transition to identify and rectify any discrepancies before patient harm occurs. Medication review is the process of evaluating current medication treatment to manage the risk and optimize the outcomes of medication treatment by detecting, solving, and preventing medication-related problems. The present study focuses on medication assessment including both medication reconciliation and review combined to clinical assessment of an individual patient.

According to a systematic review there is a need for research focusing on medication management in community settings and especially to assess the impact of medication assessment on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Home dwelling ≥65 years-old persons registered to public home care services and who

1. have had dizziness, orthostatic hypotension or have fallen or
2. use at least six medicines

Exclusion Criteria:

Home care is not responsible for patient's medication, for example due to severe chronic illness (for example severe renal insufficiency or cancer with active treatment in secondary or tertiary care).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 514 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Functional capacity IADL (Instrumental Activities of Daily Living) | at 6 months from baseline
Functional capacity ADL (Activities of daily living;KATZ) | at 6 months from baseline
Functional capacity TUG (Timed up and go) | at 6 months from baseline
Functional capacity MMSE ( Mini-mental state examination) | at 6 months from baseline
Functional capacity GDS (Geriatric Depression Scale)-15 | at 6 months from baseline

SECONDARY OUTCOMES:
Use of health care services | at 6 and 12 months from baseline
  visits to physician, hospital days and nursing care at home
Need of services delivered to home | at 6 and 12 months from baseline
Number of medicines | at 6 and 12 months from baseline
Quality of medicines | at 6 and 12 months from baseline
Cost of medicines | at 6 and 12 months from baseline
Health related quality of life assessed with EQ-5D | at 6 and 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Mäntyselkä, MD, Study Chair — Professor
Locations (5):
- Finland (5):
  - Welfare district of Forssa, Forssa
  - Selänne Basic Health Care District, Haapajärvi
  - Juva Health Care, Juva
  - City of Lahti, home care, Lahti
  - Eastern Savo Hospital District, Savonlinna

REFERENCES:
- [Derived] Auvinen K, Voutilainen A, Jyrkka J, Lonnroos E, Mantyselka P. Interprofessional medication assessment among home care patients: any impact on functioning? Results from a randomised controlled trial. BMC Geriatr. 2020 Oct 6;20(1):390. doi: 10.1186/s12877-020-01796-1. PMID 33023497